CLINICAL TRIAL: NCT06569498
Title: Neoadjuvant Transcatheter Arterial Chemoembolization Combined With Lenvatinib Plus Cadonilimab for Resectable Hepatocellular Carcinoma: A Single-Arm Phase II Clinical Trial
Brief Title: Neoadjuvant Triple Therapy for Resectable HCC
Acronym: TALENP001
Status: Recruiting | Type: Observational
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Mao-Lin Yan, Department of Hepatobiliary Pancreatic Surgery, Fujian Provincial Hospital
Other Study IDs: TALENP001
Record Dates: First submitted 2024-07-28; First posted 2024-08-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Resectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a single-arm, multi-center, prospective phase II trial aimed at evaluating the efficacy and safety of neoadjuvant therapy with transarterial chemoembolization (TACE) combined with lenvatinib and camrelizumab (triple therapy) in patients with resectable hepatocellular carcinoma (HCC). The study plans to enroll 20 patients. The primary endpoints are major pathological response (MPR) rate and safety, while the secondary endpoints are recurrence-free survival (RFS), objective response rate (ORR), R0 resection rate, and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the study and sign the informed consent form.
2. Male or female patients aged between 18 and 75 years.
3. Child-Pugh class A.
4. Indocyanine green 15-minute retention rate (ICGR-15) < 15%.
5. ECOG performance status 0-1.
6. Diagnosed with hepatocellular carcinoma (HCC) according to the "Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2022 Edition)."
7. BCLC stage A or B, with a single tumor larger than 5 cm or multiple tumors, and considered surgically resectable after multidisciplinary discussion.
8. According to RECIST 1.1 criteria, the patient has at least one measurable lesion (a measurable lesion with a long diameter ≥ 10 mm on CT/MRI scan, and the measurable lesion has not received local treatments such as radiotherapy or cryotherapy).
9. Blood routine: absolute neutrophil count ≥ 1.5 × 10^9/L, Hb ≥ 8.5 g/L, PLT ≥ 75 × 10^9/L.
10. No history of severe arrhythmia, heart failure, severe pulmonary ventilation disorders, or severe lung infections; no acute or chronic renal failure, and creatinine clearance rate > 40 mL/min.
11. Women of childbearing potential must agree to use contraception during the medication period and for 6 months after the end of medication; have a negative serum or urine pregnancy test within 7 days prior to enrollment, and must not be breastfeeding. Men must agree to use contraception during the study period and for 6 months after the end of the study.

Exclusion Criteria:

1. Tumor rupture with bleeding or suspected abdominal cavity metastasis.
2. Previous treatment with any antitumor therapies before enrollment, such as targeted drugs, PD-1/PD-L1/CTLA-4 monoclonal antibodies, surgery, TACE, FOLFOX systemic chemotherapy, radiotherapy, and Huaier granules.
3. History of allergy to lenvatinib, cadonilimab, or their components.
4. Presence of any active autoimmune disease or a history of autoimmune disease with expected recurrence (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases and syndromes); hypothyroidism treated with stable doses of thyroid replacement hormone; type 1 diabetes mellitus treated with stable doses of insulin; excluding patients with vitiligo or childhood asthma/allergies that have resolved and require no intervention in adulthood.
5. History of immunodeficiency; patients using immunosuppressive drugs or systemic corticosteroids for immunosuppressive purposes and who have continued using them within 2 weeks before signing the informed consent form.
6. Known hereditary or acquired bleeding (e.g., coagulopathy) or thrombotic tendency, such as hemophilia; currently receiving or recently (within 10 days before the start of study treatment) receiving full-dose oral or injectable anticoagulants or thrombolytics for therapeutic purposes (prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed).
7. Severe infection within 4 weeks before the first use of the study drug (CTC AE grade > 2), such as severe pneumonia requiring hospitalization, bacteremia, or infection complications; baseline chest imaging indicating active lung inflammation; symptoms and signs of infection within 2 weeks before the first use of the study drug or requiring oral or intravenous antibiotic treatment (excluding prophylactic antibiotic use).
8. Urinalysis indicating proteinuria ≥ 1+; if so, a 24-hour urine protein test is required; patients with 24-hour urine protein ≥ 1 g.
9. History of other malignancies within the past 5 years or concurrently, except for cured basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid carcinoma.
10. Patients with concomitant psychiatric disorders; history of substance abuse, alcohol, or drug addiction.
11. Pregnant or breastfeeding women.
12. Patients with significant surgical contraindications, such as renal and cardiopulmonary insufficiency, as judged by the investigator, or any other reasons deemed unsuitable for participation in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma being treated at Fujian Provincial Hospital or other centers participating in this study
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
MPR rate | Immediately after surgery
  The proportion of residual viable tumor cells in the tumor bed of the surgically resected specimen ≤10%.
Adverse events | From the initiation of medication, with recordings made whenever an adverse reaction occurs, assessed up to 12 months.
  Refer to the adverse events related to study medication, including type, incidence, and severity; severity was graded according to NCI CTCAE Version 5.0.
Operative mortality | From date of surgery, assessed up to 1 month.
  Defined as the rate of death occurring in the hospital or within 30 days of surgery.
Operative complications | From date of surgery, assessed up to 12 months.
  Defined as complications directly related to surgery and graded according to the Clavien-Dindo classification.
Reoperation rate | From date of surgery, assessed up to 12 months.
  Defined as the percentage of postoperative complications that were resolved by surgical treatment.

SECONDARY OUTCOMES:
RFS | From date of surgery until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  The time interval between the date of surgery and the first recurrence, or death from any cause.
ORR | Four weeks after the initiation of medication until the day before surgery
  The proportion of individuals whose best overall response is a complete response (CR) or partial response (PR) according to the mRECIST1.1 criteria.
R0 resection rate | Immediately after surgery
  The proportion of patients who achieve R0 resection (defined as the rate of negative margins microscopically).
OS | From date of surgery until the date of death from any cause, assessed up to 60 months.
  The time interval between the date of surgery and death from any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Fujian provincial hospital, Fuzhou, Fujian
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhongshan Hospital of Xiamen University, Xiamen, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian

IPD SHARING:
Plan to Share IPD: No